CLINICAL TRIAL: NCT02667301
Title: Investigation of Activities of Paratubal Muscles for Opening Eustachian Tube as Assessed by Simultaneous Electromyography and Tympanic Air Exchange Observations
Brief Title: Eustachian Tube Dysfunction Assessment
Acronym: ETDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stratejik Yenilikci Girisimler Ltd. (Industry)
Collaborators: Haseki Training and Research Hospital (Other); The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Murat Haluk Ozkul, Head, ENT Clinic Education and Training, Haseki Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ETDA-1
Record Dates: First submitted 2016-01-15; First posted 2016-01-28 (Estimated); Results first posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Eustachian Tube Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EMG, TAS and tympanometry (Experimental): All treatments were performed by the same group of professionals. EMG needle administration by an ENT specialist with 30+ year experience, EMG recording by a neurologist with 20+ year experience. Tympanic cavity Air exchange Sensor (TAS) recording is done by an experienced technician. The following are done to all patients:
  1. The patient is subjected to tympanometry test on the specific ear,
  2. The patient is subjected to TAS test on the specific ear while sipping water and signals from ear and nasal cavity recorded,
  3. The patient is hooked up to EMG instrument and TAS test equipment simultaneously and signals are recorded by both instruments for a duration of 150-300 seconds while the patient is at rest without sipping water. The patient is allowed to swallow during the test.
  Interventions: Device: EMG recording; Device: Tympanic Cavity Air Exchange Test; Device: Tympanometer test

INTERVENTIONS:
Device: EMG recording — 1.3X0.4 mm, sterile subdermal monopolar needle electrodes along with the same type of reference needle electrodes were inserted mTVP and mLVP muscles submucosally through the soft palate trans orally. The point of insertion for mTVP was one mm inferior and lateral of the pterygoid hamulus which is palpable at the posterior-medial of the upper alveolus. The active electrode was fully inserted horizontally into the superior belly of mTVP on the tested side. The reference electrode for mTVP was inserted into the palatine aponeurosis at one centimeter apart from the active electrode. The point of insertion for the mLVP active electrode was one centimeter medial and five mm inferior to the hamulus pterygoideus. Reference electrode of mLVP was inserted into one cm apart of medial side of the passive electrode of the mTVP at palatine aponeurosis.
  Other Names: EMG Medelec ®Synergy
Device: Tympanic Cavity Air Exchange Test — Tympanic cavity air exchange test is done by placing a sensitive pressure sensor in the ear canal and another pressure sensor on one of the nostrils. Patient is asked to to obstruct the other nostril with his/her index finger while holding the probe in place securely and asked to swallow the water during the next ten seconds. Both ear canal and nasal pressure values were simultaneously recorded on tympanic cavity air exchange sensor computer for subsequent analyses. The swallowing action triggers the ET opening and causes a momentary increase of pressure in the nasal cavity. ET opening moves the tympanic membrane which is sensed by the sensors.
  Other Names: TAS (Tympanic cavity Air exchange Sensor)
Device: Tympanometer test — Patient is subjected to tympanometry test on the specific ear and information is recorded.
  Other Names: Sonic GSI 39

SUMMARY:
The purpose of the study is to understand the exact mechanism of the activity of paratubal muscles in opening eustachian tube in patients with the functional eustachian tube and those with the eustachian tube dysfunction problem.

DETAILED DESCRIPTION:
In this study adult patients with normal and abnormal middle ears with documented tympanogram were tested to detect the Levator Veli Palatini (mLVP) and the tensor Veli Palatini (mTVP) electromyographic (EMG) activities corresponding to eustachian tube (ET) opening at rest. The subjects were mixed some with and some without ET dysfunction (ETD). Tests were conducted at an audiology unit at a tertiary care center located near at sea level, constant atmospheric pressure and temperature. Subjects are to be selected randomly with and without eustachian tube dysfunction (ETD) by using a questionnaire and evaluated with tympanometry and tympanic air exchange testing of the external ear canal for testing the ET openings. Monopolar and reference needle electrodes for each muscle were inserted transpalatally on the test side without topical anesthetics. Tympanic air exchange test is done by placing a pressure sensor into the external ear canal of the patient as well as a nasal pressure sensor for detecting ET openings during EMG recording. Information received from ear pressure and nasal pressure sensor of tympanic air exchange sensor (TAS) equipment was used for assessing the swallowing efficacy of the healthy subjects. Simultaneous correspondent recordings of the ET openings during the test as well as the electromyographic activity for the mLVP, mTVP were recorded.

ELIGIBILITY:
Inclusion criteria:

* Patients are selected from outpatients visiting Department of Otolaryngology of Haseki Hospital with a mixture of healthy Eustachian tube and with Eustachian Tube Dysfunction problem who agreed to participate in the study after being informed and signed the consent form. Questionnaire (ETDQ-7) is used for initial determination of those with and without ET dysfunction problem to include the sufficient number of patients with ETD problem in the batch.

Exclusion criteria:

* All of the subjects had an examination of the tympanic membrane, middle ear, nasal cavity and nasopharynx.
* Patients with severe septal deformities, nasal polyps and turbinate hypertrophy, adenoid and other nasopharyngeal masses were excluded.
* Patients with upper respiratory tract infections, acute otitis media, tympanosclerosis, otosclerosis and those who had previous ear surgery were not included in the study group.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided
IPD for all participants are available

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in Haseki Training and Research Hospital. An ETDQ7 questionnaire was filled out in patients who came to the Otorhinolaryngology clinic of Haseki hospital and had various ear complaints. Patients with a score of 14.5 points or greater in this quantitative test were accepted as potential "chronic eustachian dysfunction patients
Pre-assignment Details: 39 enrolled participants were excluded from the study before assignment to the group because of unreliable EMG records generating wrong electrode placement for Tensor Veli Palatini and Levator Veli Palatini muscles in the soft palate.
Groups:
- EMG, TAS and Tympanometry: All treatments were performed by the same group of professionals. EMG needle administration by an ENT specialist with 30+ year experience, EMG recording by a neurologist with 20+ year experience. Tympanic cavity Air exchange Sensor (TAS) recording is done by an experienced technician. The following are done to all patients:
  1. The patient is subjected to tympanometry test on the specific ear,
  2. The patient is subjected to TAS test on the specific ear while sipping water and signals from ear and nasal cavity recorded,
  3. The patient is hooked up to EMG instrument and TAS test equipment simultaneously and signals are recorded by both instruments for a duration of 150-300 seconds while the patient is at rest without sipping water. The patient is allowed to swallow during the test.
  Tympanometer test: Patient is subjected to tympanometry test on the specific ear and information is recorded.
Period: Overall Study
Arm/Group | EMG, TAS and Tympanometry
Started | 16
Completed | 14
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | EMG, TAS and Tympanometry
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Latency Between mLVP and mTVP Signals
Description: The time difference between mLVP and mTVP signals. This is an indication of synchronization of muscle activities.
Time Frame: Test is conducted within 60 days after enrolling the patient
Measure: Mean (Standard Deviation); unit: Time in milliseconds
Arm/Group | EMG, TAS and Tympanometry
Number analyzed (Participants) | 16
Time in milliseconds | 127.26 (61.028420946845)

2. Secondary Outcome: Amplitude in mTVP and mLVP in Microvolts
Time Frame: Test is conducted within 60 days after enrolling the patient
Measure: Mean (Standard Deviation); unit: microvolts
Groups:
- mLVP: Recorded amplitude of mLVP
- mTVP: Recorded amplitude of mTVP
Arm/Group | mLVP | mTVP
Number analyzed (Participants) | 16 | 16
microvolts | 650 (211.3315816689) | 1075 (247.71225993981)

3. Other Pre Specified Outcome: Observations About the Phase Relationship Between the Signal Pattern of mLVP, mTVP and Eustachian Dysfunction Problem
Description: Any observable relationship between the signal patterns and eustachian dysfunction problem which helps to our understanding of eustachian dysfunction problem and the electrical activity of ET muscles. Common characteristics of patients with healthy and unhealthy eustachian tube.
Time Frame: Within 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | EMG, TAS and Tympanometry
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EMG, TAS and Tympanometry (N=16)
Anxiety (Psychiatric disorders) | 1 (1) — Anxiety from procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-08-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT02667301/Prot_000.pdf